CLINICAL TRIAL: NCT02709967
Title: Cluster Randomized Trial on the Effectiveness of a Girls' Empowerment Programme on Early Childbearing, Marriage and School Dropout Among Adolescent Girls in Rural Zambia
Brief Title: Research Initiative to Support the Empowerment of Girls
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: University of Zambia (Other); Chr. Michelsen Institutt (Unknown); Norwegian School of Economics (Unknown)
Responsible Party: Principal Investigator, IFSandoey, Professor, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015/895
Record Dates: First submitted 2016-03-02; First posted 2016-03-16 (Estimated); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Pregnancy in Adolescence
MeSH Terms: interventions — Economics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Material support (Active Comparator): Writing materials
  Interventions: Other: Material support
- Economic support (Experimental): Writing materials and economic support (monthly cash transfer to girls, annual grant to guardians, and payment of school fees in grade 8 and 9).
  Interventions: Other: Material support; Other: Economic
- Combined intervention (Experimental): Writing materials, economic support (monthly cash transfer to girls, annual grant to guardians, and payment of school fees in grade 8 and 9) and community dialogue (youth club meetings, community and parent meetings)
  Interventions: Other: Material support; Other: Economic; Behavioral: Community dialogue

INTERVENTIONS:
Other: Material support — Writing materials
Other: Economic — Economic support (monthly cash transfer to girls, annual grant to guardians, and payment of school fees in grade 8 and 9)
  Arms: Combined intervention; Economic support
Behavioral: Community dialogue — Community dialogue (youth club meetings, community and parent meetings)
  Arms: Combined intervention

SUMMARY:
Background Adolescent pregnancies carry risks to the young mothers and the babies. Keeping girls in school can potentially protect girls from getting pregnant. In Zambia, 35% of young rural girls have given birth by the age of 18 years, and the pregnancy rates are particularly high among girls who are out-of-school. Approximately 50% of girls never enroll in secondary school. Widespread myths and negative social norms are barriers to adolescent girls using modern contraceptives, thus contributing to high rates of early pregnancy. However, there is little robust research from Africa on how sexual and reproductive health programmes can be delivered in a way that actually affects early marriage and pregnancy rates.

Purpose To measure the effect on early childbearing rates and basic school completion in a rural Zambian context of (1) economic support to girls and their families, and (2) combining economic support with a community intervention to enhance knowledge about sexual and reproductive health and supportive community norms

Design Cluster randomized controlled trial with three arms with clusters being rural basic schools (With grades 1-9) with surrounding communities.

Study population The participant population were girls enrolled in grade 7 in January in 2016 in rural schools in twelve study districts: Kalomo, Choma, Pemba, Monze, Mazabuka, Chikankata, Kapiri Mposhi, Kabwe, Chisamba, Chibombo, Mkushi, and Luano.

Study size A total of 4922 girls and 157 clusters were recruited, that is 999 girls and 31 clusters in the control arm and 2004 and 63 clusters in the economic support arm and 1919 girls and 63 schools in the combined intervention arms. The rationale for having different numbers of clusters was that we expected larger differences between each of the intervention arms and the control arm than between the two intervention arms themselves.

Intervention One intervention arm was offered economic support in the form of monthly cash transfers to the participating girl and her parents and payment of junior secondary school fees in 2017 and 2018. The second intervention arm was offered the same economic support combined with a community component comprising community meetings about the value of education for adolescent girls and the risks related to early childbearing, and a youth club covering comprehensive sexuality education for girls and boys (both in- and out-of-school).

DETAILED DESCRIPTION:
Background Adolescent pregnancies carry risks to the young mothers and their babies. Keeping girls in school can potentially protect girls from getting pregnant. In Zambia, 35% of young rural girls have given birth by the age of 18 years, and the pregnancy rates are particularly high among girls who are out-of-school. Approximately 50% of girls never enroll in secondary school. A number of studies have found that economic support to girls and/or their families can increase school enrolment and attendance, and three trials have found effects on postponement of childbearing and marriage. Other studies indicate that widespread myths and negative social norms are barriers to adolescent girls using modern contraceptives, thus contributing to high rates of early pregnancy. However, there is little robust research from Africa on how sexual and reproductive health programmes can be delivered in a way that actually affects early marriage and pregnancy rates.

Purpose To measure the effect on early childbearing rates and basic school completion in a rural Zambian context of (1) providing economic support to girls and their families, and (2) combining economic support with a community intervention to enhance knowledge about sexual and reproductive health and supportive community norms.

Design Cluster randomized controlled trial with three arms with clusters being rural basic schools (With grades 1-9) with surrounding communities.

Study population The participant population will be girls enrolled in grade 7 in January in 2016 in rural schools in twelve study districts: Kalomo, Choma, Pemba, Monze, Mazabuka, Chikankata, Kapiri Mposhi, Kabwe, Chisamba, Chibombo, Mkushi, and Luano.

Study size A total of 4922 girls and 157 clusters were recruited, that is 999 girls and 31 clusters in the control arm and 2004 and 63 clusters in the economic support arm and 1919 girls and 63 schools in the combined intervention arms. The rationale for having different numbers of clusters was that we expected larger differences between each of the intervention arms and the control arm than between the two intervention arms themselves.

Intervention The control group (31 schools) received writing materials. One intervention group (63 schools) was offered writing materials and economic support in the form of monthly cash transfers to the participating girl and her parents and payment of junior secondary school fees in 2017 and 2018. The second intervention group (63 schools) was offered writing materials, economic support, and a community component. The community component comprised of community meetings about the value of education for adolescent girls and the risks related to early childbearing, and a youth club covering comprehensive sexuality education for girls and boys (both in- and out-of-school).

Duration and Follow-up The duration of the trial, from recruitment to the last follow-up survey was 4.5 years. A baseline survey was conducted just after recruitment, and a final survey was conducted after approximately 4.5 years. In between there were short follow-up contacts with all the participants every six months.

Primary objectives

1. To measure the effectiveness of a combined economic and community intervention on childbearing within 8 months of the end of the intervention period
2. To measure the effectiveness of economic support alone and of a combined economic and community intervention on childbearing before the 18th birthday among girls.
3. To measure the effectiveness of economic support alone and of a combined economic and community intervention on the proportion of girls who sit for the grade 9 exam.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Enrolled in grade 7

Exclusion Criteria:

* Moved permanently away from catchment area of school

Ages: 9 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4922 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Incidence of births within 8 months of the end of the intervention | 44 months after recruitment
  Will be measured using follow up questionnaire, validated against measurement with final survey questionnaire
Incidence of births before girls' 18th birthday | 56 months after recruitment
  Will be measured using final survey questionnaire
Proportion of girls who sit for grade 9 exam | 56 months after recruitment
  Will be measured using final survey questionnaire, validated against exam register

SECONDARY OUTCOMES:
Incidence of marriage/ cohabitation before girls' 16th birthday | 56 months after recruitment
  Will be measured using final survey questionnaire
Incidence of marriage/ cohabitation before girls' 18th birthday | 56 months after recruitment
  Will be measured using final survey questionnaire
Socioeconomic inequality in incidence of marriage/ cohabitation before girls' 18th birthday | 56 months after recruitment
  Marriage/cohabitation will be measured using final survey questionnaire. We will use two measures of socioeconomic status: (i) guardian's highest level of education and (ii) household per capita consumption. Both socioeconomic measures will be categorized into tertiles of similar size.
Incidence of pregnancies among girls within 2 years of the end of the interventions | 56 months after recruitment
  Will be measured using final survey questionnaire
Incidence of births among girls within 2 years of the end of the interventions | 56 months after recruitment
  Will be measured using final survey questionnaire
Incidence of pregnancies before girls' 16th birthday | 56 months after recruitment
  Will be measured using final survey questionnaire, validated against measurement with follow-up questionnaire at 24-48 months post-recruitment
Incidence of births before girls' 16th birthday | 56 months after recruitment
  Will be measured using final survey questionnaire, validated against measurement with follow-up questionnaire at 24-48 months post-recruitment
Incidence of pregnancies before girls' 18th birthday | 56 months after recruitment
  Will be measured using final survey questionnaire
Socioeconomic inequality in incidence of births before girls' 18th birthday | 56 months after recruitment
  Births will be measured using final survey questionnaire. We will use two measures of socioeconomic status: (i) guardian's highest level of education and (ii) household per capita consumption. Both socioeconomic measures will be categorized into tertiles of similar size.
Proportion of girls enrolled in grade 8 | 12 months after recruitment
  will be measured using follow-up questionnaire, validated against school registers
Average examination scores of girls from grade 9 in English, mathematics and science | 34 months after recruitment
  will be measured using grade 9 exam results obtained from District educational boards
Proportion of girls who enrol in grade 10 | 38 months after recruitment
  will be measured using follow-up questionnaire, validated against school registers and final survey questionnaire at 56 months post-recruitment
Socioeconomic inequality in participation in grade 9 exam among girls | 56 months after recruitment
  Participation in grade 9 will be measured using final questionnaire, validated against exam register. We will use two measures of socioeconomic status: (i) guardian's highest level of education and (ii) household per capita consumption. Both socioeconomic measures will be categorized into tertiles of similar size.
Proportion currently using modern contraceptives | 32 months after recruitment
  Will be measured using final survey questionnaire
Knowledge of modern contraceptives among adolescent girls | 32 months after recruitment
  Will be measured using final survey questionnaire
Perceived community norms regarding modern contraceptive use among unmarried adolescent girls | 32 months after recruitment
  Will be measured using final survey questionnaire
Perceived community norms regarding early marriage | 32 months after recruitment
  Will be measured using final survey questionnaire
Perceived community norms regarding adolescent pregnancy | 32 months after recruitment
  Will be measured using final survey questionnaire
Perceived community norms regarding education among girls | 32 months after recruitment
  Will be measured using final survey questionnaire
Proportion of adolescent girls who have been sexually active in last 4 weeks | 32 months after recruitment
  Will be measured using final survey questionnaire
Proportion of girls currently employed or self-employed | 56 months after recruitment
  Will be measured using final survey questionnaire
School attendance of girls in grade 8 | 12 and 18 months after recruitment
  will be measured using follow-up questionnaire, validated against school registers. Attending 4 or more days per week on average will be categorized as high attendance, and less than 4 days on average will be categorized as low attendance.
School attendance of girls in grade 9 | 24 and 30 months after recruitment
  will be measured using follow-up questionnaire, validated against school registers. Attending 4 or more days per week on average will be categorized as high attendance, and less than 4 days on average will be categorized as low attendance.

CONTACTS AND LOCATIONS:
Overall Officials: Ingvild F Sandøy, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided
not yet determined

REFERENCES:
- [Derived] Mori AT, Mudenda M, Robberstad B, Johansson KA, Kampata L, Musonda P, Sandoy I. Impact of cash transfer programs on healthcare utilization and catastrophic health expenditures in rural Zambia: a cluster randomized controlled trial. Front Health Serv. 2024 Apr 29;4:1254195. doi: 10.3389/frhs.2024.1254195. eCollection 2024. PMID 38741917
- [Derived] Mori AT, Kampata L, Musonda P, Johansson KA, Robberstad B, Sandoy I. Cost-benefit and extended cost-effectiveness analysis of a comprehensive adolescent pregnancy prevention program in Zambia: study protocol for a cluster randomized controlled trial. Trials. 2017 Dec 19;18(1):604. doi: 10.1186/s13063-017-2350-4. PMID 29258591